CLINICAL TRIAL: NCT05053906
Title: Effect of Functional Endoscopic Sinus Surgery On Eustachian Tube Function in Patients With Nasal Polypi
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safia Saleh Abdellattef, Assistant lecturer, Assiut University
Other Study IDs: FESS
Record Dates: First submitted 2021-03-21; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Functional Endoscopic Sinus Surgery
MeSH Terms: interventions — Endoscopes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endoscope — effect of FESS on eustachian tube function

SUMMARY:
This study is conducted to :

Correlate the incidence of ETD with nasal polypi. To evaluate the effects of functional endoscopic sinus surgery on eustachian tube function in patients with nasal polypi

DETAILED DESCRIPTION:
Eustachian tube dysfunction (ETD) is a frequently applied diagnosis, used when abnormal ET function is believed to underlie any of a wide range of symptoms or middle ear (ME) abnormalities. Two distinct forms of the disorder are recognised, representing different ends of the spectrum of ET function: 1)obstructive ETD (OETD), in which tubal opening or patency is reduced, and 2) patulous ETD (PETD), in which the ET is too open. It has been suggested that some patients with OETD have either predominantly active dysfunction (failure of muscle-controlled opening), or passive dysfunction (failure of pressure-related opening).

There are several explanations to account for the ET dysfunction associated with nasal diseases:

* Mechanical obstruction of ET orifice may occur due to nasal mass.
* Increased secretions from seromucous glands in the pharyngeal portion of ET may accumulate and block the tube.
* Lymphatic stasis due to edema of the submucosa of the tube resulting in compromise of the lumen may produce ET dysfunction.
* Further increase in hydrostatic pressure result in the accumulation of ME fluid by transudative process.
* Tubal dysfunction may be related to deficiency of surfactant that is thought to facilitate tubal opening. It has been postulated that this material is inactivated by inflammation.

ETD symptoms will decrease post-endoscopic sinus surgery to a level comparable with a non-CRS population The use of the ETDQ-7 has the potential to enhance clinical care by highlighting the impact of ETD as well as guiding and evaluating appropriate management. Further prospective testing of

ELIGIBILITY:
Inclusion Criteria:

* Patient Who have been diagnosed to have nasal polypi Both unilateral and bilateral before doing FESS

Exclusion Criteria:

* children Patient. Patients with craniofacial abnormalities or active infection Patients with suspected nasal and nasopharyngeal tumour Patients with nasal and ear surgery

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients planned for FESS who have nasal polypi will undergo a complete history and physical examination (including otoscopy and palpation of the face and temporomandibular joints), pre-operative nasal endoscopy, computed tomography (CT) of the paranasal sinuses , completion of the Eustachian Tube Dysfunction questionnaires -7 and tempanometry. And Postoperative : nasal endoscopy, , completion of the Eustachian Tube Dysfunction questionnaires -7 and tempanometry
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The rate of Eustachian tube dysfunction with nasal polyp | 2years

REFERENCES:
- [Background] Csakanyi Z, Katona G, Konya D, Mohos F, Sziklai I. Middle ear gas pressure regulation: the relevance of mastoid obliteration. Otol Neurotol. 2014 Jul;35(6):944-53. doi: 10.1097/MAO.0000000000000282. PMID 24691503
- [Background] Ilan O, Marcus EL, Cohen Y, Farkash T, Levy R, Sasson A, Adelman C. Eustachian tube dysfunction leading to middle-ear pathology in patients on chronic mechanical ventilation. J Laryngol Otol. 2017 Sep;131(9):817-822. doi: 10.1017/S0022215117001554. Epub 2017 Jul 31. PMID 28758602